CLINICAL TRIAL: NCT04550026
Title: Cardiovascular Effects of Heated Tobacco Products (HTP)
Acronym: ISMOKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Lundbäck, MD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-03387
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Heated Tobacco Products; Microcirculation; Thrombosis; Vascular Function; Blood Markers; Microvesicles; NETs
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalation of HTP (Experimental): Inhalation of HTP for 30 minutes
  Interventions: Other: HTP inhalation
- Sham inhalation of HTP (Active Comparator): Sham usage of HTP for 30 minutes
  Interventions: Other: HTP inhalation

INTERVENTIONS:
Other: HTP inhalation — Sham inhalation for 30 minutes
  Other Names: HTP inhalation for 30 minutes

SUMMARY:
This is a human randomized controlled cross-over study where the effects of heated tobacco products (HTP) on vascular function, microcirculation and thrombosis is assessed.

DETAILED DESCRIPTION:
The World Health Organization estimates that smoking is one of the leading causes of premature death worldwide with an estimated 5-8 million lives lost annually due to tobacco usage (1).

Heated tobacco products (HTP) is a new form of tobacco products. HTP usually consists of a pod with tobacco that is mixed with glycerol which is inserted into a heating chamber. HTP is not combusted but only heated (2). Previous studies into smoking cessation with regular cigarettes and electronic cigarettes have suggested a risk for double usage instead of cessation, augmenting a nicotine addiction (3-5). There is a risk that HTP use simply enhances nicotine usage and smoking addiction.

There is limited data on the health effects of HTP. A majority of the studies available have reported conflicts of interest to manufacturers of HTP (11). It has been shown that aerosols from HTP contain toxic compounds and free radicals just as in regular cigarette smoke, albeit in lower concentrations (6-8). Furthermore, aerosols from HTP can spread in a room, enabling passive exposure (9). It has been shown that there is a decrease in harmful biomarkers in smokers that switch to HTP after 5 days of usage but also of a higher HTP consumption compared to regular smoking (12). There are few studies on effects of HTP in humans. Nabavizadeh et al has shown impaired endothelial function in rats after exposure to IQOS (10).

_____________

Subjects and criteria:

Thirty male or female occasional tobacco users (age 18-40, maximum 10 cigarettes per month or 10 pouches of snus per month) will be included. They have to be healthy, having no preexisting conditions or take any medications. All subjects will have to complete a normal health declaration.

Methods:

In randomized cross-over fashion subjects will either inhale vapor (1 puff per minute for 30 minutes, total 30 puffs) from a HTP of the brand IQOS (IQOS 3 Multi, Philip Morris AB) or perform sham-smoking of HTP. Measurements of arterial stiffness is performed previous, during and 60 minutes following exposures. Blood samples will be collected at baseline for cotinine, measurement with T-TAS, endothelial progenitor cells (EPC), NETs and extracellular vesicles (EV). Blood samples will be drawn up to 3 hours post-exposure (EPC, T-TAS,EV, NETs). Microcirculation is evaluated at baseline with skin capillaroscopy and Laser-Speckle contrast imaging (LSCI) and at 1 hour post-exposure.

Measurement of vascular function Arterial stiffness (Sphygmocor) Increased arterial stiffness is recognized as a major factor in vascular aging and a risk factor for cardiovascular disease (13). Arterial stiffness will be assessed by pulse wave analysis and pulse wave velocity.

Photopletysmography (PPG) Finger photoplethysmography is another method that provides information on the arterial bloodflow which allows measurement of pulse propagation time (PPT) (14).

Measurement of microcirculation Microcirculation will be assessed by several methods. Skin perfusion is investigated through Laser Speckle contrast Imaging , which is an optical technique for assessment of skin flux, i.e movement of circulating red blood cells. This method measures overall skin flux in superficial arterioles, capillaries and venules over wide skin areas and with a high frequency. Iontophoresis is a non-invasive method for drug application across the skin using a small electric current. Acetylcholine (ACh, Sigma-Aldrich AB, Stockholm, Sweden) and sodium nitroprusside (SNP, Hospira, Inc., Lake Forest, IL, USA), both diluted in 9% physiological sodium chloride solutions, are used to investigate endothelium-dependent and endothelium-independent microvascular reactivity, respectively. Electrode chambers (LI611 Drug Delivery Electrode, Perimed, Järfälla, Sweden) are attached to the volar side of the left forearm, avoiding hair, broken skin and visible veins, and filled with a small volume of either ACh (2%) or SNP (2%). A battery-powered iontophoresis controller (Perilont LI 760; Perimed, Järfälla, Sweden) provides a single dose of 0.02 mA for 200 seconds for drug iontophoresis. ACh is delivered using an anodal charge and SNP with a cathodal charge. LSCI (PeriCam PSI NR; Perimed, Järfälla, Sweden) is used to assess skin microvascular flux continuously before, during and 15 minutes after iontophoresis.

Skin capillaroscopy is another method for evaluating the microcirculation. A USB microscope (CapillaryScope 500 pro, Dino-Lite®) is used to visualize nail fold capillaries in the finger (preferably 4th digit of left hand). Capillaries with good optical signals, i.e. with visible red blood cell movements and plasma gaps, are chosen for examination. Capillary blood flow is registered continuously at rest, during and after one-minute arterial occlusion at the proximal phalanx of the digit with a suprasystolic cuff pressure. Calculation of capillary blood cell velocity (CBV, mm/s) is done off line and will generate following four variables: rCVB (mean CBV at rest), pCVB (peak CBV following one-minute arterial occlusion), time to peak (time (s) from release of cuff pressure to peak flow, and post-occlusive reactive hyperemia (precentral increase of CBV from rest to peak flow).

Blood pressure:

A semi-automatic oscillometric sphygmomanometer will be used to measure blood pressure and heart rate.

Blood sampling Blood samples will be drawn into test tubes containing 1/10 0.129 M sodium citrate, EDTA and serum at baseline, at 2 hour and 4 hours after exposure. Plasma is later collected after centrifugation at 2 000g for 20 min in room temperature (RT) and then frozen at -70°C until analysis.

Measurement of thrombus formation (T-TAS) T-TAS® (Total Thrombus-formation Analysis System) is a means of assessing thrombus formation during variable flow conditions using a small blood sample.

Measurement of cotinine Measurement is done to ensure adherence that subjects have not used tobacco in the last 7 days. Levels of cotinine will be measured in serum using a commercial available ELISA technique.

Measurement of EPCs The number of EPCs will be measured in whole blood by flow cytometry. EPCs are measured as CD34+ KDR+ (KDR: vascular endothelial growth factor receptor 2) double positive cells. Briefly, 20 µl of whole blood is incubated with CD34-FITC (Beckman Coulter, Brea, CA, USA) and CD309 (Becton Dickinson, Franklin Lakes, New Jersey, USA). Conjugate isotype-matched immuno-globulin (IgG1-FITC, IgG1-PE) with no reactivity against human antigens are used as a negative control. After 30 minutes of incubation in a dark environment, BD cell-fix is added to fixate the samples. Twenty thousand events of leukocytes are collected (based on classical forward scatter/side scatter (size/granularity) characteristics of blood leukocytes) and results will be presented as a number of EPC events.

Measurement of Extracellular Vesicles Plasma is thawed and centrifuged at 2000g for 20 minutes at RT. The supernatant is then re-centrifuged, at 13 000g for 2 minutes at RT. 20 µl of sample is incubated for 20 minutes in dark with phalloidin-Alexa-660 (Invitrogen, Paisley, UK), lactadherin-FITC (Haematologic Technologies, Vermont, USA), CD42a-PE (Platelet-MP (PMP), BD, Clone Alma-16), CD45-PC7 (Leukocyte-EV (LEV), Beckman Coulter, Dublin, Ireland) and CD144-APC (Endothelial-EV (EEV), AH diagnostics, Stockholm, SWE). PEVs are also labeled with CD154-PE (CD40L, abcam, Cambridge, UK) and EEVs with CD62E (E-selectin, Beckman Coulter, Dublin, Ireland). EVs are measured by flow cytometry on a Beckman Gallios instrument (CA, USA). The EV-gate is determined using Megamix beads (BioCytex, Marseille, France), which is a mix of beads of with diameters of 0.5 µm, 0.9 µm and 3.0 µm, respectively. EVs are defined as particles less than 1.0 µm in size, negative to phalloidin (in order to exclude cell membrane fragments) and positive to lactadherin. Conjugate isotype-matched immunoglobulin (IgG1-FITC, IgG1-PE, IgG1-APC and IgG1- PC7) with no reactivity against human antigens is used as a negative control to define the background noise of the cytometric analysis. The absolute number of EVs is calculated by means of the following formula: (EV counted x standard beads ⁄ L) ⁄ standard beads counted, (FlowCount, Beckman Coulter).

__________________

References

1. World Health Organization, & Others. (2019). WHO Report on the Global Tobacco Epidemic, 2019. Geneva: World Health Organization; 2019. Google Scholar.
2. Smith, M. R., Clark, B., Lüdicke, F., Schaller, J.-P., Vanscheeuwijck, P., Hoeng, J., & Peitsch, M. C. (2016). Evaluation of the Tobacco Heating System 2.2. Part 1: Description of the system and the scientific assessment program. Regulatory Toxicology and Pharmacology: RTP, 81 Suppl 2, S17-S26.
3. Lee, S., R.A. Grana, and S.A. Glantz, Electronic Cigarette Use Among Korean Adolescents: A Cross-Sectional Study of Market Penetration, Dual Use, and Relationship to Quit Attempts and Former Smoking. J Adolesc Health, 2013.
4. Caponnetto, P., et al., Impact of an electronic cigarette on smoking reduction and cessation in schizophrenic smokers: a prospective 12-month pilot study. Int J Environ Res Public Health, 2013. 10(2): p. 446-61.
5. Polosa, R., et al., Effect of an electronic nicotine delivery device (e-Cigarette) on smoking reduction and cessation: a prospective 6-month pilot study. BMC Public Health, 2011. 11: p. 786.
6. Bekki, K., Inaba, Y., Uchiyama, S., & Kunugita, N. (2017). Comparison of chemicals in mainstream smoke in heat-not-burn tobacco and combustion cigarettes. Journal of UOEH. https://doi.org/10.7888/juoeh.39.201
7. Shein, M., & Jeschke, G. (2019). Comparison of Free Radical Levels in the Aerosol from Conventional Cigarettes, Electronic Cigarettes, and Heat-Not-Burn Tobacco Products. Chemical Research in Toxicology. https://doi.org/10.1021/acs.chemrestox.9b00085
8. Ruprecht, A. A., De Marco, C., Saffari, A., Pozzi, P., Mazza, R., Veronese, C., … Boffi, R. (2017). Environmental pollution and emission factors of electronic cigarettes, heat-not-burn tobacco products, and conventional cigarettes. Aerosol Science and Technology. https://doi.org/10.1080/02786826.2017.1300231
9. Mitova, M. I., Campelos, P. B., Goujon-Ginglinger, C. G., Maeder, S., Mottier, N., Rouget, E. G. R. Tricker, A. R. (2016). Comparison of the impact of the Tobacco Heating System 2.2 and a cigarette on indoor air quality. Regulatory Toxicology and Pharmacology. https://doi.org/10.1016/j.yrtph.2016.06.005
10. Nabavizadeh, P., Liu, J., Havel, C. M., Ibrahim, S., Derakhshandeh, R., Jacob, P., & Springer, M. L. (2018). Vascular endothelial function is impaired by aerosol from a single IQOS HeatStick to the same extent as by cigarette smoke. Tobacco Control. https://doi.org/10.1136/tobaccocontrol-2018-054325
11. Simonavicius, E., McNeill, A., Shahab, L., & Brose, L. S. (2019). Heat-not-burn tobacco products: A systematic literature review. Tobacco Control. https://doi.org/10.1136/tobaccocontrol-2018-054419
12. Yuki, D., Takeshige, Y., Nakaya, K., & Futamura, Y. (2018). Assessment of the exposure to harmful and potentially harmful constituents in healthy Japanese smokers using a novel tobacco vapor product compared with conventional cigarettes and smoking abstinence. Regulatory Toxicology and Pharmacology. https://doi.org/10.1016/j.yrtph.2018.05.001
13. Mahmud, A., & Feely, J. (2003). Effect of smoking on arterial stiffness and pulse pressure amplification. Hypertension. https://doi.org/10.1161/01.HYP.0000047464.66901.60
14. Sommermeyer, D., Zou, D., Ficker, J. H., Randerath, W., Fischer, C., Penzel, T., … Grote, L. (2016). Detection of cardiovascular risk from a photoplethysmographic signal using a matching pursuit algorithm. Medical and Biological Engineering and Computing. https://doi.org/10.1007/s11517-015-1410-8
15. Mahmud, A., & Feely, J. (2003). Effect of smoking on arterial stiffness and pulse pressure amplification. Hypertension, 41(1), 183-187.

ELIGIBILITY:
Inclusion Criteria:

* Normal health declaration

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of pulmonary disease like asthma or COPD
* Any form of systemic or chronic disorder like rheumatologic or metabolic diseases. - Symptoms of infection or inflammation within 4 weeks of the study
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
microcirculation microcirculation | change from baseline and 1 hour following exposures
  Iontophoresis and laser speckle contrast imaging (LSCI),
thrombosis (total thrombus formation analysis system) | change from baseline up to 3 hour following exposures]
  T-TAS (area under the curve, flow pressure change)
arterial stiffness | change from baseline up to 3 hour following exposures]
  PWV, PWA
Microvesicles | change from baseline up to 3 hour following exposures
  microvesicles of leukocyte, endothelial and platelet origin (MVs/microliter)
NETs(neutrophil extracellular traps) | change from baseline up to 3 hours following exposures
  blood levels of H3Cit using ELISA
capillary microscopy | change from baseline to 1 hour following exposures]
  capillary blood cell velocity, CBV, mm/s
Endothelial progenitor cells | change from baseline up to 3 hours following exposures
  EPC

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Jernberg, MD, Prof, Study Director — Karolinska Institutet
Locations (1):
- Institutionen för kliniska vetenskaper, Danderyds sjukhus, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No